CLINICAL TRIAL: NCT02674451
Title: Remote Ischemic Preconditioning to Prevent Contrast-induced Nephropathy in Patients With Stable and Unstable Coronary Disease Undergoing Coronary Angiography.
Brief Title: Remote Ischemic Preconditioning to Prevent Contrast Nephropathy
Acronym: RIPC-CIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00036762
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC (Active Comparator): Participants will receive remote ischemic preconditioning within one hour of coronary angiography. This involves blood pressure cuff inflation to 200mmHG for three-5 minute periods, each separated by 5 minute intervals.
  Interventions: Procedure: Remote ischemic preconditioning
- Controls (Sham Comparator): Participants will have routine blood pressure measurements will be obtained.
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Blood pressure cuff inflation to 200 mmHG for three 5-minute periods each separated by 5 minute intervals within 1 hour of planned coronary angiography.

SUMMARY:
Contrast-medium induced nephropathy (CIN) is a frequent and devastating complication of coronary angiography, occurring in 10-50% of cases. As would be expected, the incidence of CIN is much higher in patients with underlying renal dysfunction. Multiple trials have found CIN to be an independent predictor of prolonged hospitalization and both 30 day and 1 year mortality in patients with coronary artery disease. Intravenous contrast dye is felt to cause renal ischemia as the mechanism of injury. Unfortunately, despite the significant morbidity and mortality with CIN, there are few therapeutic interventions to reduce the risk with the exception of hydration and high dose statin therapy. Recently, remote ischemic preconditioning (RIPC), a process of inducing transient arm ischemia by inflating a blood pressure cuff to 200 mmHg for 3 repetitive 5 minute cycles, leads to a systemic cytoprotective response and ultimately reduces ischemic renal injury, myocardial injury, and even cerebral injury following coronary bypass grafting. While there is significant data supporting the role of RIPC in reducing systemic ischemic injury in surgical patients, there is only one small trial studying RIPC in patient's undergoing coronary angiography. The investigators hypothesize that RIPC will reduce the incidence of contrast-induced nephropathy in patients with baseline renal dysfunction undergoing coronary angiography for stable or unstable coronary artery disease.

DETAILED DESCRIPTION:
Contrast-medium induced nephropathy (CIN) is a frequent and devastating complication of coronary angiography, occurring in 10-50% of cases dependent on individual risk factors (JACC 2004; 44:1393). Multiple trials have found CIN to be an independent predictor of prolonged hospitalization and both 30 day and 1 year mortality in patients with coronary artery disease (Clin Res Cardiol 2009;98:765, JACC 2004:44:1780, Ann Int Med 2009;150:170, JACC 2008; 51: 1419). The largest retrospective study of over 16,000 hospitalized patients exposed to iodinated contrast found an in-hospital mortality rate of 34% in subjects developing CIN versus 7% in matched control subjects (JAMA 1996;275:1489). Despite the incidence of CIN and the deleterious outcomes, few therapies exist to prevent CIN other than hydration and withdraw of nephrotoxic medications prior to coronary angiography.

Remote ischemic preconditioning (RIPC) is a protective response resulting from transient episodes of ischemia, followed by reperfusion, to vascular beds remote from the organ which will undergo the prolonged ischemic insult. Studies in humans indicate that RIPC decreases cardiac enzyme release, clinical events, and improves mortality in patients undergoing elective coronary bypass surgery (Circulation 2009;119:820; Lancet 2007;370:575, Lancet 2013; 382: 597). In addition to the cardio-protective effects of RIPC, a small, single center randomized trial showed a reduction in the incidence of contrast-medium induced nephropathy of approximately 30% in patients receiving RIPC prior to elective coronary angiography compared to a control population (Circulation 2012; 126:296). RIPC was safely performed in all of these studies by inflating a blood pressure cuff to supra-systolic levels (200mmHg) for 3 five minute episodes separated by 5 minutes of reperfusion.

RIPC is a well-tolerated, easily administered mechanism that may reduce the incidence of contrast-mediated nephropathy. However, additional and larger trials are needed to validate the use of RIPC in both elective and urgent coronary angiography in patients at risk for contrast-medicated nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography for stable or unstable coronary artery disease
* eGFR less than or equal to 60 mL/min/1.73 m2

Exclusion Criteria:

* Subjects with known upper extremity vascular disease
* Subjects with systolic blood pressure differential of 10 mmHg or higher in the upper extremities
* End stage renal disease on peritoneal or hemodialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 48 hours after contrast administration
  Increase in serum creatinine greater than or equal to 0.05 mg/dL or a relative increase of greater than or equal to 25% of baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Schulman, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No